CLINICAL TRIAL: NCT03521180
Title: Model Development, Clinical Study to Evaluate Gluten Challenge on Immune Responses in Subjects With Celiac Disease.
Brief Title: A Study to Evaluate Gluten Challenge on Immune Responses in Subjects With Celiac Disease
Status: Completed | Type: Observational
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Other Study IDs: NDS-CP-002; U1111-1208-7879 (Registry Identifier: WHO)
Record Dates: First submitted 2018-04-16; First posted 2018-05-11 (Actual); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Celiac Disease
Keywords: Celiac Disease; Gluten; Immune Response; Challenge
MeSH Terms: conditions — Celiac Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — The ICF relates that biospecimens will be retained at the central laboratory or another secure storage facility. It does make it clear samples will be destroyed after 5 years. Or that subjects can withdraw and have their samples destroyed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with Celiac Disease: Group 1 will start the gluten challenge with 4 slices of white bread once daily for 3 days. Blood will be taken at pre-specified time points for up to 9 days following the start of gluten challenge for biomarker analyses.
  Based on data from the first 5 subjects, the 2nd group of 5 subjects may: 1) not be needed if the objectives are met; 2) receive gluten at increased quantity (not to exceed 6 slices of bread once daily for 3 days) or have biomarker samples collected at adjusted time points; 3) same as the first 5 subjects; 4) reducing the duration of gluten free diet for a minimum of 3 months instead of 6 month for the Inclusion Criteria # 5;5) subjects may be re-enrolled once.
  The same applies to the 3rd group of subjects. A notification will be provided to the clinical study site for detailed changes.

SUMMARY:
This is a model development, open label, no therapeutic treatment, three sequential group, short term-gluten challenge study in subjects with celiac disease. Immune responses are evaluated following gluten challenge.

Approximately fifteen subjects with celiac disease will be enrolled in up to three sequential groups (5 subjects per group).

ELIGIBILITY:
Inclusion Criteria:

Subjects must satisfy the following criteria to be enrolled in the study:

1. Male and female subjects of any race between 18 to 65 years of age (inclusive) at the time of signing the informed consent form (ICF).
2. Must understand and voluntarily sign an ICF prior to any study-related assessments/procedures being conducted.
3. Must be able to communicate with the investigator, understand and comply with the requirements of the study, and agree to adhere to restrictions and examination schedules.
4. Documented diagnosis of celiac disease ≥ 6 months before study entry, based on American College of Gastroenterology 2013 guideline on celiac disease diagnosis and management. The confirmation of a diagnosis of CD should be based on a combination of findings from the medical history, physical examination, serology, and upper endoscopy with histological analysis of multiple biopsies of the duodenum.

   1. A positive biopsy consistent with celiac disease. Every effort should be made to obtain the biopsy report to support the diagnosis of CD. Prospective subjects should not undergo biopsy for the sole purpose for participating in this trial. And
   2. A documented positive gluten-specific serology to tissue transglutaminase (tTG), endomysial antibodies (EMA), and/or gliadin-derived peptides (GDP).
5. Group 1 subjects must have been following a gluten-free diet for ≥ 6 months before study entry and have been in remission based on self-reporting and must have negative IgA antibodies to tTG at screening. For Group 2 and 3 the gluten free diet duration may be reduced to a minimum of 3 months. Notification of the changes for Group 2 and 3 will be provided to the site(s).
6. Subjects must have HLA DQ2.5 (i.e., DQA1*05/DQB1*02).
7. No clinically significant abnormal laboratory test results other than those related to celiac disease as determined by the investigator.
8. At the screening visit, must be afebrile, with supine systolic BP: 90 to 140 mmHg, supine diastolic BP: 50 to 90 mmHg, and pulse rate: 40 to 110 bpm. Eligibility criteria for vital signs performed on Day 0 (or Day 1 pre-gluten challenge) will be at the discretion of the Investigator. In the opinion of the Investigator, subjects with hypertension controlled with a concomitant medication will be allowed in the study.
9. Must have a normal or clinically acceptable 12-lead ECG.
10. Female subject must have a negative pregnancy test at screening and on Day 0 (or Day 1 pre-gluten challenge).
11. Subject must be willing and able to adhere to the study visit schedule and other protocol requirements.

Exclusion Criteria:

The presence of any of the following will exclude a subject from enrollment:

1. Any significant medical condition, laboratory abnormality, or psychiatric illness, Type 1 diabetes, other than celiac disease, that would prevent the subject from participating in the study.
2. Any condition which places the subject at unacceptable risk if he were to participate in the study, or confounds the ability to interpret data from the study.
3. Use of any prescribed systemic immune modulator medication within 30 days of the first bread administration.
4. The use of prescribed and over-the-counter non-steroidal anti-inflammatory drugs (NSAID) within 14 days of the first bread administration.
5. Exposure to an investigational drug (new chemical entity) within 30 days prior to the first bread administration or 5 half-lives of that investigational drug, if known (whichever is longer).
6. Donated blood or plasma within 8 weeks before the first bread administration to a blood bank or blood donation center.
7. History of drug abuse (as defined by the current version of the Diagnostic and Statistical Manual [DSM]) within 2 years before dosing, or a positive drug screen reflecting consumption of illicit drugs. For states in which marijuana is legal; prior use of marijuana may be acceptable as long as the screening drug screen is negative. Subjects may be re-screened in case the drug screen tests positive for marijuana. Subjects must refrain from the use of marijuana 2 weeks prior to screening until the end of study.
8. History of alcohol abuse (as defined by the current version of the DSM) within 2 years before screening, or a positive alcohol screen.
9. Known to have hepatitis, or known to be a carrier of the hepatitis B surface antigen (HBsAg) or hepatitis C antibody (HCV Ab), or have a positive result to the test for human immunodeficiency virus (HIV) antibodies at screening.
10. Any condition that confounds the ability to interpret data from the study.
11. Subjects with a history of hypersensitivity or anaphylaxis to gluten.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: A total of approximately 15 subjects (male or female) with celiac disease will be enrolled. Subjects must be positive for the HLA-DQ2.5+ haplotype. The disease should be well controlled through gluten-free diet. They must have followed a strict gluten free diet prior to screening with no symptoms that would suggest accidental gluten ingestion during that time.
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2018-05-11 (Actual); Primary Completion 2019-07-18 (Actual); Study Completion 2019-07-18 (Actual)

PRIMARY OUTCOMES:
Gut-homing, activated, CD8+ αβ T cells and γδ T cells in PBMC | Approximately 10 days
  The number of gut-homing, activated, CD8+ αβ T cells and γδ T cells in PBMC will be reported separately by flow cytometry .
Evaluation of Gliadin reactive T cell measures- PBMC (peripheral blood mononuclear cells) by Flow Cytometry | Approximately 10 days
  Gliadin specific T cells will be evaluated by flow cytometry using fluorescently labelled HLA-gliadin tetramers that selectively bind to gliadin-specific T-cells.
Gliadin reactive T cell measures- PBMC (peripheral blood mononuclear cells) by ELISPOT | approximately 10 days
  Gliadin specific T cells will be evaluated using Enzyme-linked immunospot (ELISPOT) which measure the number of cells secreting cytokine in response to gliadin binding.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Ye, PhD, Study Director — Celgene
Locations (2):
- United States (2):
  - Covance, Dallas, Texas
  - Virginia Mason Medical Center, Seattle, Washington